CLINICAL TRIAL: NCT06467799
Title: Neoadjuvant Hepatic Arterial Infusion Chemotherapy Plus Tislelizumab Combined With Adjuvant Tislelizumab in Preventing Postoperative Recurrence for High-risk Hepatocellular Carcinoma: a Prospective, Single-arm, Phase II Clinical Study
Brief Title: Neoadjuvant HAIC and PD-1 Plus Adjuvant PD-1 for High-risk Recurrent HCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Chen Min-Shan, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B2024-211-01
Record Dates: First submitted 2024-06-13; First posted 2024-06-21 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Hepatocellular Carcinoma; Beyond Milan Criteria
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental arm (Experimental): Two cycles of FOLFOX-HAIC combined with tislelizumab as neoadjuvant therapy, followed by surgical resection and four cycles of adjuvant tislelizumab.
  Interventions: Drug: Neoadjuvant HAIC and PD-1 Plus Adjuvant PD-1

INTERVENTIONS:
Drug: Neoadjuvant HAIC and PD-1 Plus Adjuvant PD-1 — Patients will first receive two cycles of FOLFOX-HAIC combined with tislelizumab as neoadjuvant therapy, with a 3-week interval between cycles. Two weeks after completing the neoadjuvant therapy, imaging assessments will be conducted to evaluate treatment efficacy and surgical feasibility. Surgical resection should be performed within two weeks following the imaging assessment. Four weeks post-resection, patients will undergo a follow-up evaluation to assess postoperative recovery and determine the presence of any residual tumor. If no residual or recurrent tumor is detected, adjuvant therapy with tislelizumab will commence (every three weeks, for a total of four cycles).

SUMMARY:
Surgical resection is the primary curative treatment for patients with hepatocellular carcinoma (HCC), with a 5-year overall survival rate of 60-80% post-surgery. Therefore, guidelines recommend surgical resection as the first-line choice for early to mid-stage HCC (CNLC stages IA-IIA or BCLC stages A/B) patients with well liver reserve function. However, the high postoperative recurrence rate is the main factor limiting long-term survival in HCC patients, with literature reporting recurrence rates exceeding 70%. Among these, half of the patients experience recurrence within two years post-surgery, imposing a heavy burden on patients' physical and mental health as well as on societal medical resources. Adopting effective treatment to improve surgical curability and reduce postoperative recurrence rates is one of the current research hotspots.

Recent studies from the investigators' center indicate that hepatic arterial infusion chemotherapy (HAIC) and immunotherapy can provide definite efficacy for patients with advanced HCC, extending their survival time. Mechanistically, chemotherapy and immunotherapy have synergistic effects: tumor cell necrosis induced by chemotherapy can promote immune activation, while cytokines and neutralizing antibodies secreted by immune cells can enhance the toxicity of chemotherapeutic drugs.

Therefore, this study aims to conduct a prospective, single-arm, phase II clinical study, targeting HCC patients with high-risk recurrence factors, to evaluate whether neoadjuvant HAIC combined with a PD-1 monoclonal antibody (Tislelizumab) followed by adjuvant Tislelizumab post-surgery can reduce postoperative recurrence rates in HCC patients. The primary endpoint is the 1-year recurrence-free survival (RFS) rate post-surgery, while secondary endpoints include the objective response rate (ORR) of neoadjuvant therapy, the incidence of perioperative complications, the incidence of treatment-related adverse events, overall survival (OS) time, pathological complete response (pCR) rate of neoadjuvant therapy, and major pathological response (MPR) of neoadjuvant therapy. The investigators aim to comprehensively assess the efficacy and safety of neoadjuvant HAIC plus PD-1 and adjuvant PD-1 in the perioperative treatment of HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed and untreated hepatocellular carcinoma (clinical diagnostic criteria based on the " Chinese Guidelines for the Diagnosis and Treatment of Hepatocellular Carcinoma (2024 Edition) " formulated by the National Health Commission of China and the Barcelona Clinic Liver Cancer (BCLC) strategy for prognosis prediction and treatment recommendation of the European Association for the Study of the Liver (EASL));
2. Tumor staging: beyond Milan criteria (single tumor >5 cm, or 2-3 tumors with the largest diameter >3 cm), resectable CNLC stage Ib/IIa hepatocellular carcinoma;
3. No tumor thrombus, distant metastasis, or lymph node metastasis;
4. Normal liver volume ≥ 700 cc, estimated residual liver volume >40% after resection;
5. Patient KPS ≥ 90;
6. Liver function Child-Pugh class A;
7. Estimated survival of more than 6 months;
8. Function of important organs meets the following requirements: white blood cells ≥ 4.0×10^9/l, neutrophils ≥ 1.5×10^9/l, platelets ≥ 80.0×10^9/l, hemoglobin ≥ 90 g/l; serum albumin ≥ 2.8 g/dl; total bilirubin ≤ 1.5 × ULN, ALT/AST/ALP ≤ 2.5 × ULN; serum creatinine ≤ 1.5 × ULN or creatinine clearance rate > 60 mL/min; no severe organic diseases;
9. The subject must be able to understand and voluntarily sign a written informed consent form, and must sign the informed consent form prior to any specific procedure of the study, agreeing to comply with the medication and postoperative follow-up requirements as designed in this study.

Exclusion Criteria:

1. Combined with severe impairment of functions of other important organs such as heart, lungs, and kidneys; active infections other than viral hepatitis or other serious comorbid conditions, making the patient unable to tolerate treatment;
2. Contraindications to surgical resection and immunotherapy;
3. History of other malignant tumors;
4. Combined with immunological diseases or other conditions requiring long-term steroid treatment;
5. Known or suspected allergy to the study drug or any drugs administered in connection with this trial;
6. History of organ transplantation;
7. Pregnant or breastfeeding women;
8. Other factors that may affect patient enrollment and assessment outcomes;
9. Refusal to follow-up according to the requirements set by the study protocol, and refusal to sign the informed consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
recurrence free survival, RFS | From date of treatment beginning until the date of first documented tumor recurrence or date of death from any cause, whichever came first, assessed up to 1 years
  RFS is defined as the time from treatment to post-resection tumor recurrence or death from any cause.

SECONDARY OUTCOMES:
objective response rate，ORR | From date of neoadjuvant treatment beginning until the date of neoadjuvant treatment completion, up to 1 year.
  The ratio of patients achieving the best efficacy of neoadjuvant therapy, including complete response (CR) and partial response (PR), to all patients.
pathological complete response，pCR | From date of neoadjuvant treatment beginning until the date of surgical resection completion, , up to 1 year.
  The ratio of patients with no viable tumor cells in the pathology after resection to all patients undergoing surgical resection.
overall survival, OS | From date of treatment beginning until the date of death from any cause, assessed up to 1 years.
  OS is defined as the time from randomization to death from any cause.
perioperative complication rate | The period from the start of surgery to the patient's discharge from hospital, up to 1 year.
  Perioperative complication includes intraoperative complications such as bleeding and transfusion, extensive adhesions, diaphragm resection, prolonged surgery time, etc., as well as postoperative complications such as bleeding, infection, bile leakage, liver dysfunction, etc.
Incidence of adverse events (safety ) | From date of neoadjuvant treatment beginning until the date of adjuvant treatment completion, up to 2 year.
  Treatment-related adverse events are evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (CTCAE 5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Yaojun Zhang, MD, PHD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China